CLINICAL TRIAL: NCT00410098
Title: The Influence of Bikram Yoga (39 Degree Celsius Heat and 60% Humidity) on Basic Lung Function Tests,Bronchial Challenges and Pulmonary-Heart Endurance in Young Asthmatic Adults.
Brief Title: Bikram Yoga and Asthma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: bikramasthma-HMO-CTIL
Record Dates: First submitted 2006-12-10; First posted 2006-12-12 (Estimated); Last update posted 2006-12-12 (Estimated); Status verified 2006-12

CONDITIONS: Asthmatics
Keywords: asthma; yoga; heat; humidity; bikram
MeSH Terms: conditions — Asthma

INTERVENTIONS:
Behavioral: Bikram Yoga

SUMMARY:
Cold and dry air induce exercise induced asthma. Yoga training may improve lung function tests. Bikram Yoga (heat 39 degree Celsius and humidity 60%)training may improve both lung function tests and bronchial hyperreactivity (to exercise and adenosine 5'monophosphate).

DETAILED DESCRIPTION:
15 young adults with exercise induced asthma and 10 healthy young adults will participate in 2 months taining of Bikram Yoga in Tel Aviv. They will perform sessions of 90 minutes training at least 5 times a week. Lung function tests, bronchial challenges (exercise and AMP) and progressive exercise test will be performed before and after the 2 month training at Hadassah University Hospital in Jerusalem in the asthmatic patients. Healthy adults will perform only lung function tsts and progressive exercise before and after training.

ELIGIBILITY:
Inclusion Criteria:

* controlled asthma
* age 18-30 years

Exclusion Criteria:

* heart,
* hypertension,
* kidney disease,
* chronic lung disease,
* oxygen dependence

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-06

PRIMARY OUTCOMES:
prevent exercise induced asthma and improve lung function tests

CONTACTS AND LOCATIONS:
Overall Officials: Avraham AVITAL, MD, Prof, Principal Investigator — Hadassah Medical Organization